CLINICAL TRIAL: NCT05375396
Title: Assessment of Colonization of Dairy Free Probiotic Bacterium Streptococcus Salivarius From Lozenges to the Oral Cavity
Brief Title: Microbial Colonization of Dairy Free Oral Probiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: John Hale (Industry)
Responsible Party: Sponsor-Investigator, John Hale, Chief Technology Officer, BLIS Technologies Limited
Organization: BLIS Technologies Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BLTCT2022/4
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Microbial Colonization
Keywords: Streptococcus salivarius M18; dairy free; allergen free; probiotic; microbial colonization; oral probiotic; chewable tablet
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Probiotic Streptococcus salivarius M18 lozenges Probiotics dairy free Streptococcus salivarius M18 lozenges
Who Masked: Participant, Investigator
Masking Description: A staff member not part of the study group will be assigned to distribute blinded samples. The participant or the investigators will not be aware of the dose groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Streptococcus salivarius M18 lozenges (Active Comparator): Streptococcus salivarius M18 lozenges containing dairy based Streptococcus salivarius M18
  Interventions: Dietary Supplement: Streptococcus salivarius M18 lozenges
- Streptococcus salivarius M18 dairy free lozenges (Active Comparator): Streptococcus salivarius M18 lozenges containing dairy free Streptococcus salivarius M18
  Interventions: Dietary Supplement: Streptococcus salivarius M18 dairy free lozenges

INTERVENTIONS:
Dietary Supplement: Streptococcus salivarius M18 lozenges — In this study, a lozenge formulation containing dairy based S. salivarius M18 will be evaluated for its potential of delivering probiotic Streptococcus salivarius M18 to the oral cavity.
  Arms: Streptococcus salivarius M18 lozenges
Dietary Supplement: Streptococcus salivarius M18 dairy free lozenges — In this study, a lozenge formulation containing dairy free S. salivarius M18 will be evaluated for its potential of delivering probiotic Streptococcus salivarius M18 to the oral cavity.
  Arms: Streptococcus salivarius M18 dairy free lozenges

SUMMARY:
The aim of this study is to evaluate the colonization efficacy of probiotic lozenges containing dairy and dairy free probiotic Streptococcus salivarius M18, in healthy adults

DETAILED DESCRIPTION:
This is a double-blind, randomized controlled colonization pilot study with no cross over to evaluate the colonization efficacy of two different lozenges containing either dairy or dairy free probiotic bacteria Streptococcus salivarius M18.

Participants will be randomly assigned to one of the 2 groups consuming probiotic lozenge containing dairy free Streptococcus salivarius M18 or dairy based Streptococcus salivarius M18 over a seven day period. Saliva samples will be collected at predetermined time points pre and post intervention. Colonization efficacy will be determined by enumerating the probiotic in the saliva samples using standard microbiological techniques.

ELIGIBILITY:
Inclusion criteria:

Male or Female 18y - 80y age

1. In general good health 18 - 80 years of age.
2. Practice good oral hygiene.

Exclusion criteria:

1. Have a history of autoimmune disease or are immunocompromised.
2. Are on concurrent antibiotic therapy or regular antibiotic use within last 1 week
3. History of allergy (e.g. dairy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in microbial colonization of S. salivarius M18 from Day 0 (baseline) to 1 hour | 1 hour post intervention
  Study will determine the change in microbial colonization efficacy of dairy based Streptococcus salivarius M18 in a Lozenge format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization of S. salivarius M18 from Day 0 (baseline) to 8 hours | 8 hour post intervention
  Study will determine the change in microbial colonization efficacy of dairy based Streptococcus salivarius M18 in a Lozenge format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization of S. salivarius M18 from Day 0 (baseline) to 24 hours | 24 hours post intervention
  Study will determine the change in microbial colonization efficacy of dairy based Streptococcus salivarius M18 in a Lozenge format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization of S. salivarius M18 from Day 0 (baseline) to 48hours | 48 hours post intervention
  Study will determine the change in microbial colonization efficacy of dairy based Streptococcus salivarius M18 in a Lozenge format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization of dairy free S. salivarius M18 from Day 0 (baseline) to 1 hour | 1 hour post intervention
  Study will determine the change in microbial colonization efficacy of dairy based Streptococcus salivarius M18 in a Lozenge format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization of dairy free S. salivarius M18 from Day 0 (baseline) to 8 hour | 8 hour post intervention
  Study will determine the change in microbial colonization efficacy of dairy based Streptococcus salivarius M18 in a Lozenge format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization of dairy free S. salivarius M18 from Day 0 (baseline) to 24 hour | 24 hour post intervention
  Study will determine the change in microbial colonization efficacy of dairy based Streptococcus salivarius M18 in a Lozenge format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization of dairy free S. salivarius M18 from Day 0 (baseline) to 48 hour | 48 hour post intervention
  Study will determine the change in microbial colonization efficacy of dairy based Streptococcus salivarius M18 in a Lozenge format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).

CONTACTS AND LOCATIONS:
Overall Officials: John D D Hale, PhD, Study Director — Blis Technologies Ltd; Rohit Jain, PhD, Principal Investigator — Blis Technologies Ltd, Dunedin, New Zealand; John R Tagg, PhD, Study Director — Blis Technologies Ltd, Dunedin, New Zealand
Locations (1):
- Blis Technologies Ltd, Dunedin, Otago, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Data and information included in the Protocol and Clinical Study Report will be shared to other researchers and/or in publications in due course.
Supporting Information: Study Protocol, CSR
Time Frame: Study report 3 months after the completion of the study
Access Criteria: Summary study report will be shared by Principal Investigator upon request if not published in public literature

REFERENCES:
- [Background] Di Pierro F, Zanvit A, Nobili P, Risso P, Fornaini C. Cariogram outcome after 90 days of oral treatment with Streptococcus salivarius M18 in children at high risk for dental caries: results of a randomized, controlled study. Clin Cosmet Investig Dent. 2015 Oct 3;7:107-13. doi: 10.2147/CCIDE.S93066. eCollection 2015. PMID 26491371
- [Background] Bardellini E, Amadori F, Gobbi E, Ferri A, Conti G, Majorana A. Does Streptococcus Salivarius Strain M18 Assumption Make Black Stains Disappear in Children? Oral Health Prev Dent. 2020 Apr 3;18(2):161-164. doi: 10.3290/j.ohpd.a43359. PMID 32099975
- [Background] Burton JP, Wescombe PA, Macklaim JM, Chai MH, Macdonald K, Hale JD, Tagg J, Reid G, Gloor GB, Cadieux PA. Persistence of the oral probiotic Streptococcus salivarius M18 is dose dependent and megaplasmid transfer can augment their bacteriocin production and adhesion characteristics. PLoS One. 2013 Jun 13;8(6):e65991. doi: 10.1371/journal.pone.0065991. Print 2013. PMID 23785463
- [Background] Burton JP, Drummond BK, Chilcott CN, Tagg JR, Thomson WM, Hale JDF, Wescombe PA. Influence of the probiotic Streptococcus salivarius strain M18 on indices of dental health in children: a randomized double-blind, placebo-controlled trial. J Med Microbiol. 2013 Jun;62(Pt 6):875-884. doi: 10.1099/jmm.0.056663-0. Epub 2013 Feb 28. PMID 23449874